CLINICAL TRIAL: NCT04360746
Title: The Influence of Clinical Pharmacist on the Quality of Drug Prescribing and Rehabilitation Outcomes in Post-acute Hip Fractured Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, AVITAL HERSHKOVITZ, Head of Rehabilitation Department D, 'Beit Rivka' Geriatric Rehabilitation Center, Rabin Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 0832-19-RMC
Record Dates: First submitted 2020-04-16; First posted 2020-04-24 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Hip Fractures; Clinical Pharmacists; Rehabilitation Outcome
MeSH Terms: conditions — Hip Fractures | interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical pharmacist intervention group (Active Comparator): all hip fractured patients admitted to D1 subunit in "Beit rivka" geriatric rehabilitation center. This group will get a clinical pharmacist review of their medication and a pharmaceutical counseling to the medical staff in the first few days of admission (1-5 days post admission)
  Interventions: Other: Pharmaceutical intervention; Other: Rehabilitation
- control group (Other): The control group will include all hip fractured patients admitted to D2 subunit in "Beit rivka" geriatric rehabilitation center. This group will not receive any pharmacist intervention during their rehabilitation.
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Pharmaceutical intervention — Pharmaceutical intervention will include a complete medication review by a clinical pharmacist with the following process: medication reconciliation, medication indication and dosage check, medication effectiveness and appropriateness assessment, drug-drug or drug-disease interactions check, medication duplications check, length and cost of treatment evaluation. The pharmacist will use the following tools: Medication appropriateness index (MAI), ACB (Anticholinergic cognitive burden) score and the using the assessment of underutilization (AOU) index.
  Arms: Clinical pharmacist intervention group
Other: Rehabilitation — A multidisciplinary team provided medical, nursing, physical, occupational, and social work interventions. Rehabilitation care include: (a) individual physical therapy (PT), 2 to 3 times a week; (b) 30 to 40 min of PT in an adapted fitness room, aerobic training on a treadmill with and without partial weight support and stationary bicycles, 2 to 3 times a week ; (c) 30 to 40 min of virtual reality training by performing challenging functional tasks, 2 times a week and (d) 30 to 45 min of individual occupational therapy (OT), cognitive evaluation and stimulation, safety education, and learning to use assistive devices, 3 times a week.

SUMMARY:
The influence of clinical pharmacist on various drug related outcomes was reported in different healthcare setting including the community, long term care and during acute hospitalization. Nevertheless, data on the influence of clinical pharmacist intervention on the quality of drug prescribing and rehabilitation outcomes in post-acute hip fractured patients is scarce.

The aims of the current study are to evaluate the contribution of a clinical pharmacist on the appropriateness of drug prescribing among post-acute geriatric hip fractured patients and to investigate whether this involvement can improve rehabilitation outcomes.

The investigators hypothesis is that early review of geriatric hip fractured patients medical record by a clinical pharmacist will improve the appropriateness of drug treatment and the rehabilitation outcomes among this population.

DETAILED DESCRIPTION:
An Open label randomized prospective study of elderly patients (65 years old and above) admitted for rehabilitation after hip fracture. All study participants will be admitted in the same geriatric-rehabilitation department specialized in the rehabilitation of geriatric patients after hip fracture ("D" ward). This department is divided into 2 subunits (D1 and D2) with the same patient population but a different medical and nursing staff.

Randomization in this study will be based upon the admission subunit. The intervention group will include all hip fractured patients admitted to D1 subunit. This group will get a clinical pharmacist review of their medication and a pharmaceutical counseling to the medical staff in the first few days of admission (1-5 days post admission). The control group will include all hip fractured patients admitted to D2 subunit. This group will not receive any pharmacist intervention during their rehabilitation, unless the pharmacist will be asked directly to review a patient medical record by the medical or nursing staff. In this case the specific patient will be excluded from the study.

Pharmaceutical intervention will include a complete medication review by a clinical pharmacist with the following process: medication reconciliation, medication indication and dosage check, medication effectiveness and appropriateness assessment, drug-drug or drug-disease interactions check, medication duplications check, length and cost of treatment evaluation.

The pharmacist will use the following tools:

Medication appropriateness evaluation Medication appropriateness will be evaluated based upon the MAI (medication appropriateness index) score - an implicit (judgment-based) outcome measure. The MAI is a measure of prescribing appropriateness that assesses ten elements of prescribing: indication, effectiveness, dose, correct directions, practical directions, drug-drug interactions, drug-disease interactions, duplication, duration, and cost. Although based on implicit criteria, the index has operational definitions and explicit instructions, which standardize the rating process. Each medication can get a score between 0-18, with a higher score indicating inappropriateness of more drug elements. The ratings generate a weighted score that serves as a summary measure of prescribing appropriateness.

The clinical pharmacist will calculate the MAI score upon admission and discharge for each study participant.

Anticholinergic drug burden Anticholinergic drug burden will be assessed by a common anticholinergic drug scale. The medical literature describes several anticholinergic drug scales. Most of those scales were built by experts in order to generate an anticholinergic burden for a specific patient based upon his current drug treatment. Evaluation of the anticholinergic burden may predict the risk for an anticholinergic side effect in that patient.

the ACB (Anticholinergic cognitive burden) score will determine the anticholinergic burden for each patient. The ACB score was developed in order to evaluate the cognitive effects of anticholinergic medications. The tool gives points for each medication based on an ordinal scale. Each medication can get the following score: 0 = no potential for anticholinergic effect, 1 = slight anticholinergic effects, based on Evidence from in vitro data that chemical entity has antagonist activity at muscarinic receptor, 2 = moderate anticholinergic effects, based on evidence from literature, prescriber's information, or expert opinion of clinical anticholinergic effect, 3 = strong anticholinergic effects, based on evidence from literature, expert opinion, or prescribers information that medication may cause delirium.

The total ACB score will be calculated upon admission and discharge for each patient.

Underuse of medications Underuse of medications refers to the omission of a drug when there is a clear indication and no contraindications. The evaluation of underuse will be through a medication reconciliation process and by using the assessment of underutilization (AOU) index.

In the process of medication reconciliation the pharmacist will compare the current patient drug regimen to the recommended medications in the general hospital discharge letter and to the drugs prescribed/dispensed in the community. The purpose of this process is to trace any medication that was unintentionally omitted from the patient current drug list.

Drug Underutilizion will be assessed by the AOU tool. This instrument is intended for the evaluation of medications that should have been prescribed by a health care provider but were omitted. The pharmacist will review the medical file of each patient in search for any omission of a needed drug for an established active disease/condition.

A needed drug is defined as a drug that is indicated or recommended based on current practice guidelines or evidence available.

The study will involve pharmacist review of patient electronic medical records in order to collect the following data for each patient: the MAI and ACB at admission and discharge, the number of drugs added or stopped during the rehabilitation period, demographic data, functional level including pre-rehabilitation functional levels, cognitive function (via the mini-mental status exam) and clinical data including the metabolic state (admission albumin level), chronic diseases.

Likewise, other operation related factors will be collected, including: type of fracture, operation latency period, rehabilitation latency period and rehabilitation length of stay (LOS).

the rehabilitation outcomes for each patient will be register including the FIM score at admission and discharge, motor FIM , MRFS scores and the destination of the patient at the end of the rehabilitation period.

The same data for the control group will be collected retrospectively at the end of the study period.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patient (65 years of older) who were admitted for rehabilitation after hip fracture at "D" ward in beit rivka post-acute geriatric center.

Exclusion Criteria:

* Patient that did not complete the rehabilitation period due the following causes: death, acute care hospitalization or severe medical deterioration.
* In the case of D2 sub unit hospitalized patient - any request by the sub unit medical or nursing staff for pharmacist consultation/intervention.

Ages: 65 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Summated Medication Appropriateness Index (MAI) score | Admission (baseline value) and at discharge (approximately 5 weeks post admission)
  The change from admission to discharge in the summated medication appropriateness index score. Each medication can get a score between 0-18, with a higher score indicating inappropriateness of more drug elements.
Anticholinergic Cognitive Burden (ACB) score | Admission (baseline value) and at discharge (approximately 5 weeks post admission)
  The change from admission to discharge in the anticholinergic cognitive burden score. Each medication can get a score between 0-3, with a higher score indicating a higher anticholinergic burden.
The change in medication discrepancy | Admission (baseline value) and at discharge (approximately 5 weeks post admission)
  The number of medication discrepancy and underuse of drugs
The change in overused drugs | Admission (baseline value) and at discharge (approximately 5 weeks post admission)
  The number of overused or misused drugs
The change in Functional Independence measure (FIM) score | Admission (baseline value) and at discharge (approximately 5 weeks post admission)
  The change from admission to discharge in the Functional Independence measure score. the score is calculated for each patient and can be between 18-126, with a higher score indicating a better functional independence status.
The change in motor functional independence measure (mFIM) | Admission (baseline value) and at discharge (approximately 5 weeks post admission)
  The change from admission to discharge in motor functional independence measure score. the score is calculated for each patient and can be between 18-91, with a higher score indicating a better motor functional independence status.
The change in Montebello Rehabilitation Factor Score (MRFS) | Admission (baseline value) and at discharge (approximately 5 weeks post admission)
  The relative functional gain (motor functional independence measure effectiveness) achieved on the motor functional independence measure score. The Montebello Rehabilitation Factor Score (MRFS) is calculated as the motor functional independence measure score change (discharge score minus admission score) divided by the motor functional independence measure maximum score (a score of 91) minus the motor functional independence measure admission score. The Montebello Rehabilitation Factor Score can be between -80 to 100 with a higher score indicating a better motor functional independence measure effectiveness (a higher relative functional gain during rehabilitation).
LOS (Length Of Stay) | Through study completion, an average of 1 year
  Length of rehabilitation center stay

CONTACTS AND LOCATIONS:
Locations (1):
- Beit Rivka geriatric rehabilitation center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boparai MK, Korc-Grodzicki B. Prescribing for older adults. Mt Sinai J Med. 2011 Jul-Aug;78(4):613-26. doi: 10.1002/msj.20278. PMID 21748749
- [Background] Spinewine A, Fialova D, Byrne S. The role of the pharmacist in optimizing pharmacotherapy in older people. Drugs Aging. 2012 Jun 1;29(6):495-510. doi: 10.2165/11631720-000000000-00000. PMID 22642783
- [Background] Walsh KA, O'Riordan D, Kearney PM, Timmons S, Byrne S. Improving the appropriateness of prescribing in older patients: a systematic review and meta-analysis of pharmacists' interventions in secondary care. Age Ageing. 2016 Mar;45(2):201-9. doi: 10.1093/ageing/afv190. Epub 2016 Jan 10. PMID 26755524
- [Background] Geller AI, Nopkhun W, Dows-Martinez MN, Strasser DC. Polypharmacy and the role of physical medicine and rehabilitation. PM R. 2012 Mar;4(3):198-219. doi: 10.1016/j.pmrj.2012.02.012. PMID 22443958
- [Background] Perez T, Moriarty F, Wallace E, McDowell R, Redmond P, Fahey T. Prevalence of potentially inappropriate prescribing in older people in primary care and its association with hospital admission: longitudinal study. BMJ. 2018 Nov 14;363:k4524. doi: 10.1136/bmj.k4524. PMID 30429122
- [Background] Iaboni A, Rawson K, Burkett C, Lenze EJ, Flint AJ. Potentially Inappropriate Medications and the Time to Full Functional Recovery After Hip Fracture. Drugs Aging. 2017 Sep;34(9):723-728. doi: 10.1007/s40266-017-0482-6. PMID 28776209
- [Background] Kragh Ekstam A, Elmstahl S. Do fall-risk-increasing drugs have an impact on mortality in older hip fracture patients? A population-based cohort study. Clin Interv Aging. 2016 Apr 29;11:489-96. doi: 10.2147/CIA.S101832. eCollection 2016. PMID 27199553
- [Background] Lee JK, Alshehri S, Kutbi HI, Martin JR. Optimizing pharmacotherapy in elderly patients: the role of pharmacists. Integr Pharm Res Pract. 2015 Aug 11;4:101-111. doi: 10.2147/IPRP.S70404. eCollection 2015. PMID 29354524
- [Background] Gillespie U, Alassaad A, Hammarlund-Udenaes M, Morlin C, Henrohn D, Bertilsson M, Melhus H. Effects of pharmacists' interventions on appropriateness of prescribing and evaluation of the instruments' (MAI, STOPP and STARTs') ability to predict hospitalization--analyses from a randomized controlled trial. PLoS One. 2013 May 17;8(5):e62401. doi: 10.1371/journal.pone.0062401. Print 2013. PMID 23690938
- [Background] Viktil KK, Blix HS. The impact of clinical pharmacists on drug-related problems and clinical outcomes. Basic Clin Pharmacol Toxicol. 2008 Mar;102(3):275-80. doi: 10.1111/j.1742-7843.2007.00206.x. Epub 2008 Jan 30. PMID 18248511
- [Background] Lee JK, Slack MK, Martin J, Ehrman C, Chisholm-Burns M. Geriatric patient care by U.S. pharmacists in healthcare teams: systematic review and meta-analyses. J Am Geriatr Soc. 2013 Jul;61(7):1119-27. doi: 10.1111/jgs.12323. Epub 2013 Jun 24. PMID 23796001
- [Background] Hanlon JT, Schmader KE, Samsa GP, Weinberger M, Uttech KM, Lewis IK, Cohen HJ, Feussner JR. A method for assessing drug therapy appropriateness. J Clin Epidemiol. 1992 Oct;45(10):1045-51. doi: 10.1016/0895-4356(92)90144-c. PMID 1474400
- [Background] Samsa GP, Hanlon JT, Schmader KE, Weinberger M, Clipp EC, Uttech KM, Lewis IK, Landsman PB, Cohen HJ. A summated score for the medication appropriateness index: development and assessment of clinimetric properties including content validity. J Clin Epidemiol. 1994 Aug;47(8):891-6. doi: 10.1016/0895-4356(94)90192-9. PMID 7730892
- [Background] Somers A, Mallet L, van der Cammen T, Robays H, Petrovic M. Applicability of an adapted medication appropriateness index for detection of drug-related problems in geriatric inpatients. Am J Geriatr Pharmacother. 2012 Apr;10(2):101-9. doi: 10.1016/j.amjopharm.2012.01.003. Epub 2012 Feb 1. PMID 22304791
- [Background] Spinewine A, Schmader KE, Barber N, Hughes C, Lapane KL, Swine C, Hanlon JT. Appropriate prescribing in elderly people: how well can it be measured and optimised? Lancet. 2007 Jul 14;370(9582):173-184. doi: 10.1016/S0140-6736(07)61091-5. PMID 17630041
- [Background] Salahudeen MS, Duffull SB, Nishtala PS. Anticholinergic burden quantified by anticholinergic risk scales and adverse outcomes in older people: a systematic review. BMC Geriatr. 2015 Mar 25;15:31. doi: 10.1186/s12877-015-0029-9. PMID 25879993
- [Background] Ottenbacher KJ, Mann WC, Granger CV, Tomita M, Hurren D, Charvat B. Inter-rater agreement and stability of functional assessment in the community-based elderly. Arch Phys Med Rehabil. 1994 Dec;75(12):1297-301. PMID 7993167
- [Background] Granger CV, Hamilton BB. The Uniform Data System for Medical Rehabilitation report of first admissions for 1992. Am J Phys Med Rehabil. 1994 Feb;73(1):51-5. No abstract available. PMID 8305182
- [Background] Heruti RJ, Lusky A, Barell V, Ohry A, Adunsky A. Cognitive status at admission: does it affect the rehabilitation outcome of elderly patients with hip fracture? Arch Phys Med Rehabil. 1999 Apr;80(4):432-6. doi: 10.1016/s0003-9993(99)90281-2. PMID 10206606
- [Background] Rolland Y, Pillard F, Lauwers-Cances V, Busquere F, Vellas B, Lafont C. Rehabilitation outcome of elderly patients with hip fracture and cognitive impairment. Disabil Rehabil. 2004 Apr 8;26(7):425-31. doi: 10.1080/09638280410001663148. PMID 15204479
- [Background] Cornu P, Steurbaut S, Leysen T, De Baere E, Ligneel C, Mets T, Dupont AG. Effect of medication reconciliation at hospital admission on medication discrepancies during hospitalization and at discharge for geriatric patients. Ann Pharmacother. 2012 Apr;46(4):484-94. doi: 10.1345/aph.1Q594. Epub 2012 Mar 13. PMID 22414793
- [Background] Bulloch MN, Olin JL. Instruments for evaluating medication use and prescribing in older adults. J Am Pharm Assoc (2003). 2014 Sep-Oct;54(5):530-7. doi: 10.1331/JAPhA.2014.13244. PMID 25216883
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Spinewine A, Swine C, Dhillon S, Lambert P, Nachega JB, Wilmotte L, Tulkens PM. Effect of a collaborative approach on the quality of prescribing for geriatric inpatients: a randomized, controlled trial. J Am Geriatr Soc. 2007 May;55(5):658-65. doi: 10.1111/j.1532-5415.2007.01132.x. PMID 17493184